CLINICAL TRIAL: NCT06448546
Title: Investigating the Role of the Gut Microbiome in Huntington's Disease
Brief Title: Gut Microbiomes in HD
Status: Recruiting | Type: Observational
Sponsor: University of Central Florida (Other)
Collaborators: University of South Florida (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00006833
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Huntington Disease
Keywords: Huntington Disease; HD; Gut Microbiome
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control: Patients who are not diagnosed with HD
- Experimental Group 1: Underweight HD patients
- Experimental Group 2: Overweight HD patients

SUMMARY:
The purpose of this study is to find out if there is a connection between the naturally occurring bacteria in our bodies and the progression of Huntington disease. The investigators are trying to determine if patients who are diagnosed with adult-onset HD and who exhibit a rapid rate of disease progression have unique populations of bacteria in their gut as compared to patients with slower progression.

DETAILED DESCRIPTION:
Two of the most common non-neurological features of Huntington disease (HD) are progressive weight loss and metabolic dysfunction. However, a small proportion of HD patients are pathologically overweight, despite having similar CAG repeat lengths as pathologically underweight patients. The investigators hypothesize this spectrum of weight abnormalities may be caused by HD-related metabolic dysfunction.

Pathological weight loss is recapitulated in transgenic HD model mice expressing fragments of human huntingtin (HTT), either transgenically3,4 or knocked-in to a portion of the mouse HD homolog (Hdh) gene5. Conversely, pathological weight gain is recapitulated in transgenic HD model mice expressing full-length human HTT either along with the full complement of Hdh6,7 or in Hdh-null backgrounds8,9.

In Hdh-null background transgenic HD model mice, which are pathologically overweight, circadian feeding is disrupted, despite maintenance of naturally nocturnal circadian activity. Interestingly, circadian feeding patterns are restored by suppression of brain HTT (unpublished Dr. Amber Southwell), suggesting that HTT plays a role in circadian feeding regulation. Furthermore, when circadian feeding patterns are artificially restored with scheduled feeding, striatal HTT is temporarily suppressed, while metabolic markers and body weight are normalized (unpublished Dr. Amber Southwell). Together, this demonstrates that HTT is involved in gut-brain feedback, but since HTT suppression during scheduled feedings is transient, while metabolic effects are lasting, HTT is likely not the master regulator of this feedback loop. Instead, the gut microbiome may influence this pathway, possibly contributing to the onset and/or progression of HD.

ELIGIBILITY:
* Inclusion Criteria:

  * 18 years or older
  * Provide informed consent
  * Able to read and speak English
  * Agree to comply with study procedures
* Inclusion criteria for the control group include:

  * CAG repeat length ≤ 26.
  * BMI 18.5-24.9
* Inclusion criteria for experimental group 1 include:

  * BMI < 18.5 (underweight) or significant, involuntary weight loss within the past 12 months.
  * CAG repeat length 40 - 59.
  * Documentation of the Clinical Diagnosis of HD with a high level of certainty (>99% confidence) using the validated Unified Huntington's Disease Rating Scale (UHDRS).
  * Stage I-III on the Functional Assessment component of the UHDRS
* Inclusion criteria for experimental group 2 include:

  * BMI > 25.0 (overweight - obesity) or BMI ≤ 25.0 with significant, unexplained weight gain within the past 12 months
  * CAG repeat length 40 - 59.
  * Documentation of the Clinical Diagnosis of HD with a high level of certainty (>99% confidence) using the validated UHDRS.
  * Stage I-III on the Functional Assessment component of the UHDRS
* Exclusion Criteria:

  * CAG repeat length ≥ 60 to exclude participants with juvenile onset HD.
  * CAG repeat length 36 - 39 to exclude participants with reduced penetrance. As this is a pilot study, we are primarily interested in participants with typical HD characteristics.
  * UHDRS Functional Capacity stage ≥ 4 to exclude late-stage HD patients who may be institutionalized and receive nutrition through a feeding tube.
  * Use of any of the following drugs within the last 6 months:

    * System antibiotics, antifungals, antivirals, or anti-parasitics (intravenous, intramuscular, or oral)
    * Corticosteroids (intravenous, intramuscular, oral, nasal, or inhaled)
    * Cytokines
    * Methotrexate, immunosuppressive cytotoxic agents, or chemotherapy
    * Commercial probiotics ≥ 100 million CFU (fermented foods, yogurts, and other homeopathic probiotics and prebiotics do not apply)
  * Use of topical antibiotics or topical steroids within the last 7 days
  * History of active, uncontrolled gastrointestinal disorders or diseases, including:

    * Inflammatory bowel disease
    * Ulcerative colitis
    * Crohn's disease
    * Irritable bowel syndrome
    * Infectious gastroenteritis, colitis, or gastritis
    * Clostridium difficile or Helicobacter pylori infection
    * Persistent or chronic constipation or diarrhea
  * Acute illness with or without fever at time of sample collection
  * Positive for HIV, hepatitis B, or hepatitis C
  * Confirmed or suspected immunodeficient condition/state
  * Major surgery of the GI tract, excluding cholecystectomy and appendectomy
  * Unstable dietary history within the past month, such as elimination or significant increase of a major food group in the diet
  * Recent history of chronic, excessive alcohol consumption
  * Travel outside of the United States within the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study aims to recruit approximately 36 adult participants: 12 for the control group (who do not have the HD gene mutation), 12 for experimental group 1 (underweight HD patients), and 12 for experimental group 2 (overweight HD patients). There may be some variation in participant number depending on recruitment success. Experimental group 1 will target underweight HD patients and experimental group 2 will target normal to overweight HD patients.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
To quantify relative abundance of entire gut microbiomes in people using Metagenomic analysis | 5 years
  Metagenomic analysis via 16S ribosomal RNA (rRNA) gene sequencing will be performed on HD and control stool samples to identify HD-associated changes in microbe abundance at the genus level.

SECONDARY OUTCOMES:
To quantify relative abundance of candidate microbes in HD and control gut using quantitative PCR. | 5 years
  Using primers specific for microbes responsible for microbiota-derived metabolites that are altered in HD plasma as well as candidate microbes identified through aim 1, quantitative PCR (qPCR) will be used for quantifying relative abundance within the gut at the species level.

CONTACTS AND LOCATIONS:
Overall Officials: Amber Southwell, PhD, Principal Investigator — University of Central Florida
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No